CLINICAL TRIAL: NCT02547493
Title: Comparison of Humoral Response to Conjugate Pneumococcal Vaccine and Polysaccharide Pneumococcal Vaccine in Rheumatoid Arthritis (RA) Patients Treated With Abatacept
Brief Title: Vaccination Against Pneumococcal in Naïve Abatacept Rheumatoid Arthritis Patients
Acronym: VACINA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9419
Record Dates: First submitted 2015-09-07; First posted 2015-09-11 (Estimated); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Vaccination against Pneumococcal; Naïve Abatacept patients
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Pneumococcal Vaccines; 13-valent pneumococcal vaccine; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pneumococcal polysaccharide vaccine (Active Comparator): Patients are vaccinated vith Peumo23/Pneumovax on the first day. Abatacept started on frst day.
  Interventions: Biological: pneumococcal polysaccharide vaccine; Drug: Abatacept
- pneumococcal conjugate vaccine (Active Comparator): Patients are vaccinated with Prevenar13 on the first day, and with Pneumo23/Pneumovax two months later.
  Abatacept started on frst day.
  Interventions: Biological: pneumococcal conjugate vaccine; Drug: Abatacept

INTERVENTIONS:
Biological: pneumococcal polysaccharide vaccine — Vaccination with PPSV on first day. NB : PPSV vaccine Pneumo23 has been replaced in September 2017 by the equivalent vaccine Pneumovax because of the stop of commercialization of Pneumo23 in France by the pharmaceutical company.
  Other Names: Pneumo23/Pneumovax
  Arms: pneumococcal polysaccharide vaccine
Biological: pneumococcal conjugate vaccine — Patients are vaccinated with Prevenar13 on the first day, and with Pneumo23/Pneumovax two months later.
  Other Names: Prevenar13
  Arms: pneumococcal conjugate vaccine
Drug: Abatacept — Abatacept started on frst day
  Other Names: Orencia

SUMMARY:
Is pneumococcal conjugate vaccine (which induces a T-dependent humoral response) more efficient than pneumococcal polysaccharide vaccine (which induces a T-independent humoral response) in RA patients treated with abatacept, biotherapy targeting T-cells? The investigator propose to conduct a prospective, multicenter (11 centers), randomized, open-label study.

The patients are going to be randomized in 2 groups: patients of the first group will be vaccinated with the polysaccharide pneumococcal vaccine (Pneumo23®/Pneumovax®) whereas patients of the second group will be vaccinated with conjugate pneumococcal vaccine (Prevenar13®).

DETAILED DESCRIPTION:
The study population will be all the RA patients between 18 and 85 years with instauration of a treatment by sub-cutaneous abatacept in association with methotrexate who agreed to participate to the study.

At the time of their inclusion, patients will be randomized for receiving either pneumococcal polysaccharide vaccine (PPSV) or pneumococcal conjugate vaccine (PCV).

The primary endpoint will be evaluated at one month after vaccination. The total of follow-up will be of 12 months.

For the patients of the group PCV, the prime-boost strategy will be applied in order to be in accordance with the current French recommendation and a revaccination at 2 months after the initial vaccine will be realized with PPSV.

ELIGIBILITY:
Inclusion Criteria:

* RA according to American College of Rheumatology (ACR)/European League Against rheumatism (EULAR) 2010 criteria
* Disease Activity Score (DAS) 28 ≥ 3.2
* Initiation of a treatment by sub-cutaneous abatacept in combination with methotrexate (MTX), whatever treatment they were receiving before (apart from rituximab (RTX) in the last year)
* Patient has signed study consent form

Exclusion Criteria:

* age < 18 or > 85 year
* dementia
* patients subjects to legal protection measures
* Corticosteroids ≥ 10mg/d the day of inclusion
* Patient who had a pneumococcal vaccination in the previous 3 years
* Last pneumococcal vaccination < 3 year
* rituximab in the last year
* History of anaphylactic response to a vaccination
* Contraindications to abatacept or methotrexate
* Pregnancy or pregnancy wish
* Breast feeding
* Patient who currently abuse drugs or alcohol
* Subject who have received any live vaccines within 3 months of the anticipated first dose of study medication.
* Subject who have receive any vaccine within 1 month of the anticipated first dose of the study medication and for all the duration of the study
* Patient with contraindication to intramuscular injections
* Subject with respiratory insufficiency
* Subject at risk for Tuberculosis.
* Blood transfusion within the 3 months previous to the study and for all the duration of the study.
* Concomitant biologic disease-modifying antirheumatic drug (DMARD)
* Within 4 weeks of receiving treatment with any investigational drug.
* Patient positive for hepatitis B surface antigen
* Patient who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-03 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Humoral response comparison after vaccination (number of patient with at least a two-fold increase of the antibody titer for at least 3 of the 5 serotypes of interest : 1,3 14, 7F, 19A) | 1 month after vaccination
  To compare the rate of responders, at one month after vaccination, between patients vaccinated with PCV and patient vaccinated with PPSV.

SECONDARY OUTCOMES:
Side Effect frequency (number of side effect at each patient's visit for both groups) | 1, 2,6 ans 12 months after inclusion
  Comparison of the frequency of side effects between the 2 groups at 1, 2, 6 and 12 months
Prime boost strategy efficacity evaluation (number of responder in the PCV group) | 6 months after inclusion
  Calculation of the rate of responders, in the PCV group, at 4 month after re-vaccination by a dose of PPSV
Long term immune response after vaccination | 6 and 12 months after vaccination
  Comparison between the 2 groups of the rate of responders at 6 and 12 months after vaccination
Comparison between the 2 groups of the opsonophagocytosis activity of the antibodies produced | 1, 2, 6 and 12 months after vaccination
  Comparison between the 2 groups of the opsonophagocytic titers (OPA) at 1, 2, 6 and 12 months after vaccination
Pneumococcal vaccination predictive factor identification | 12 month after last patient inclusion
  Analysis of the collected date to search for predictive factors of immune response after pneumococcal vaccination by comparison of the rates of responders within each group, according to age, gender, RA activity, MTX dosage, corticosteroid, dosage, therapeutical history

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Morel, MD PhD, Principal Investigator — CHRU de Montpellier
Locations (11):
- France (10):
  - CHRU de Montpellier, Montpellier, Hérault
  - CHU Nord, Amiens
  - CHU Pellegrin, Bordeaux
  - CHU Montpied, Clermont-Ferrand
  - CHU Bicêtre, Le Kremlin-Bicêtre
  - CHRU Roger Salengro, Lille
  - CHU Carémeau, Nîmes
  - CHU Orléans, Orléans
  - CHU La pitié salpétriere, Paris
  - CHU Hautepierre, Strasbourg
- CHPG Monaco, Monaco, Monaco